CLINICAL TRIAL: NCT00567619
Title: LIFE NIS, GERD-Patients - Evaluation of Burden of Disease Determined by GERD Impact Scale (GIS)
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: NIS-GAT-NEX-2007/1
Record Dates: First submitted 2007-09-20; First posted 2007-12-05 (Estimated); Last update posted 2008-02-18 (Estimated); Status verified 2008-02

CONDITIONS: GERD
Keywords: GERD; NIS
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Evaluate burden of disease in Patients with newly occurred upper GI symptoms related to GERD (symptom frequency & severity, QoL, lifestyle modifications, self-medication) - baseline data according to GERD impact scale presenting to specialists, especially internists

- Evaluate effect of treatment with a acid suppressive therapy on these parameters: looking for improvement of symptom burden and quality of life according to the GERD impact sca

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly occured upper GI symptoms related to GERD

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 900
Dates: Start 2007-07

CONTACTS AND LOCATIONS:
Overall Officials: Not required for Study, Study Chair — Not required for this study
Locations (1):
- Research Site, Vienna, Austria